CLINICAL TRIAL: NCT00591916
Title: New Treatment for Donor Sites
Acronym: Donors
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Donor site material (scarlet red ) came back on the market, therefore new treatements for donor sites was not needed.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-388
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Burn
Keywords: burn; donor site; grafting; scar
MeSH Terms: conditions — Burns; Cicatrix | interventions — Scarlet Red; Hyaluronic Acid; Thrombin; Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Microbial Nanocellulose (NC), an inert material produced by Acetobacter xylinum is one of three drug interventions the patient will be randomized to receive. One of the three drugs will be placed on a patient donor site immediately after harvesting skin while the patient is in surgery.
  Interventions: Drug: Application of donor site dressing [scarlet red, Microbial Nanocellulose (NC), or hyaluronan and thrombin (HT)]; Procedure: Blood sample; Procedure: Biopsy
- 2 (Experimental): fine mesh gauze impregnated with hyaluronan and thrombin (HT) is one of three drug interventions the patient will be randomized to receive. One of the three drugs will be placed on a patient donor site immediately after harvesting skin while the patient is in surgery.
  Interventions: Drug: Application of donor site dressing [scarlet red, Microbial Nanocellulose (NC), or hyaluronan and thrombin (HT)]; Procedure: Blood sample; Procedure: Biopsy
- 3 (Active Comparator): Scarlet Red is one of three drug interventions the patient will be randomized to receive. One of the three drugs will be placed on a patient donor site immediately after harvesting skin while the patient is in surgery.
  Interventions: Drug: Application of donor site dressing [scarlet red, Microbial Nanocellulose (NC), or hyaluronan and thrombin (HT)]; Procedure: Blood sample; Procedure: Biopsy

INTERVENTIONS:
Drug: Application of donor site dressing [scarlet red, Microbial Nanocellulose (NC), or hyaluronan and thrombin (HT)] — Application of donor site dressing: scarlet red, Microbial Nanocellulose (NC), or hyaluronan and thrombin (HT).
Procedure: Blood sample — Obtain blood specimen at surgery donor site harvest, 14 days post surgery and 6 months post surgery
Procedure: Biopsy — Tissue biopsy of donor site treated area at admission, wound healing and 2-6 months post burn.

SUMMARY:
Primary research questions/Purpose of the Research.

1. Determine the short term (epidermal regeneration, reduction of pain, infections and length of stay) and long term (scarring, long term recovery, and cost of treatment) outcomes of Microbial Nanocellulose (NC) and fine mesh gauze impregnated with hyaluronan and thrombin (HT).
2. Determine if donor site treatment with NC and HT is as safe as the use of Scarlet Red ointment dressing.

   b. Describe the importance of the knowledge that you expect to gain from the research.

   To find a donor site dressing that has outcomes equal or better than that of scarlet red.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-90 years.
* Any patient admitted to the hospital with burn injury requiring grafting and a donor site.

Exclusion Criteria:

* Patient with severe burn injuries expected to die.

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
epidermal regeneration (donor site healing) | Days 3-14 post surgery

SECONDARY OUTCOMES:
Infection | Days 0-21 post surgery
reduction in pain of donor site | Day 0-21 post surgery
Scarring | Day 7 post surgery to 2 years post surgery
Costs | Admission post burn injury to 2 years post burn injury

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas